CLINICAL TRIAL: NCT06247345
Title: First in Human, Phase Ia/Ib Study for Safety, Tolerability, Pharmacokinetics, and Clinical Activity Evaluation of ADEL-Y01 in Healthy Participants and in Participants With Mild Cognitive Impairment Due to Alzheimer's Disease or Mild Alzheimer's Disease
Brief Title: A Phase Ia/Ib, First-in-human (FIH) Study for Safety, Tolerability, Pharmacokinetics (PK), and Clinical Activity Evaluation of ADEL-Y01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alzheimer's Disease Expert Lab (ADEL), Inc. (Industry)
Collaborators: Oscotec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADEL_OSCO_Y01_P101
Record Dates: First submitted 2024-01-31; First posted 2024-02-07 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Dementia; Cognitive Dysfunction; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Cognition Disorders; Tau MTBR; Disease Modifying Treatments; Monoclonal antibodies (mAbs)
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Cognition Disorders

STUDY DESIGN:
Intervention Model Description: 5 cohort in Single Ascending Dose (SAD) in healthy participants and 3 cohort in Multiple Ascending Dose (MAD) in participants with mild cognitive impairment (MCI) due to Alzheimer's Disease (AD) and mild AD
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- SAD Cohort 1: ADEL Y-01 antibody at a dose of 2.5mg/Kg (Active Comparator): This arm represents the group receiving ADEL Y-01 antibody at a dose of 2.5mg/Kg in SAD cohort 1.
  Interventions: Drug: ADEL-Y01 - healty participants
- SAD Cohort 1: Placebo at a dose of 2.5mg/Kg (Placebo Comparator): This arm represents the group receiving placebo at a dose of 2.5mg/Kg in SAD cohort 1.
  Interventions: Drug: Placebo - Healthy Participants
- SAD Cohort 2: ADEL Y-01 antibody at a dose of 7.5mg/Kg (Active Comparator): This arm represents the group receiving ADEL Y-01 antibody at a dose of 7.5 mg/Kg in SAD cohort 2.
  Interventions: Drug: ADEL-Y01 - healty participants
- SAD Cohort 2: Placebo at a dose of 7.5mg/Kg (Placebo Comparator): This arm represents the group receiving placebo at a dose of 7.5mg/Kg in SAD cohort 2.
  Interventions: Drug: Placebo - Healthy Participants
- SAD Cohort 3: ADEL Y-01 antibody at a dose of 20mg/Kg (Active Comparator): This arm represents the group receiving ADEL Y-01 antibody at a dose of 20mg/Kg in SAD cohort 3.
  Interventions: Drug: ADEL-Y01 - healty participants
- SAD Cohort 3: Placebo at a dose of 20mg/Kg (Placebo Comparator): This arm represents the group receiving placebo at a dose of 20mg/Kg in SAD cohort 3.
  Interventions: Drug: Placebo - Healthy Participants
- SAD Cohort 4: ADEL Y-01 antibody at a dose of 50mg/Kg (Active Comparator): This arm represents the group receiving ADEL Y-01 antibody at a dose of 50mg/Kg in SAD cohort 4.
  Interventions: Drug: ADEL-Y01 - healty participants
- SAD Cohort 4: Placebo at a dose of 50mg/Kg (Placebo Comparator): This arm represents the group receiving placebo at a dose of 50mg/Kg in SAD cohort 4.
  Interventions: Drug: Placebo - Healthy Participants
- SAD Cohort 5: ADEL Y-01 antibody at a dose of 100mg/Kg (Active Comparator): This arm represents the group receiving ADEL Y-01 antibody at a dose of 100mg/Kg in SAD cohort 5.
  Interventions: Drug: ADEL-Y01 - healty participants
- SAD Cohort 5: Placebo at a dose of 100mg/Kg (Placebo Comparator): This arm represents the group receiving placebo at a dose of 100mg/Kg in SAD cohort 5.
  Interventions: Drug: Placebo - Healthy Participants
- MAD Cohort 1: ADEL Y-01 antibody at a dose of 7.5mg/Kg (Active Comparator): This arm represents the group receiving ADEL Y-01 antibody at a dose of 7.5 mg/Kg in MAD cohort 1.
  Interventions: Drug: ADEL-Y01 - MCI/AD
- MAD Cohort 1: Placebo at a dose of 7.5mg/Kg (Placebo Comparator): This arm represents the group receiving placebo at a dose of 7.5mg/Kg in MAD cohort 1.
  Interventions: Drug: Placebo - MCI/AD
- MAD Cohort 2: ADEL Y-01 antibody at a dose of 20mg/Kg (Active Comparator): This arm represents the group receiving ADEL Y-01 antibody at a dose of 20mg/Kg in MAD cohort 2.
  Interventions: Drug: ADEL-Y01 - MCI/AD
- MAD Cohort 2: Placebo at a dose of 20mg/Kg (Placebo Comparator): This arm represents the group receiving placebo at a dose of 20mg/Kg in MAD cohort 2.
  Interventions: Drug: Placebo - MCI/AD
- MAD Cohort 3: ADEL Y-01 antibody at a dose of 50mg/Kg (Active Comparator): This arm represents the group receiving ADEL Y-01 antibody at a dose of 50mg/Kg in MAD cohort 3.
  Interventions: Drug: ADEL-Y01 - MCI/AD
- MAD Cohort 3: Placebo at a dose of 50mg/Kg (Placebo Comparator): This arm represents the group receiving placebo at a dose of 50mg/Kg in MAD cohort 3.
  Interventions: Drug: Placebo - MCI/AD

INTERVENTIONS:
Drug: ADEL-Y01 - healty participants — In our Part 1 clinical trial, we plan to enroll up to 40 healthy participants, aged 18 to 65, to test the safety and tolerability of ADEL-Y01. The study is divided into 5 cohorts, each with 8 participants, where 6 receive a single dose of ADEL-Y01. Screening is done 28 days prior, followed by randomization and dosing. Participants undergo initial assessments until Day 4 and additional safety and PK evaluations over 12 weeks. Starting at 2.5 mg/kg, the ADEL-Y01 dose may increase up to 100 mg/kg based on Safety Review Committee assessments, ensuring a detailed evaluation of the drug's safety.
  Arms: SAD Cohort 1: ADEL Y-01 antibody at a dose of 2.5mg/Kg; SAD Cohort 2: ADEL Y-01 antibody at a dose of 7.5mg/Kg; SAD Cohort 3: ADEL Y-01 antibody at a dose of 20mg/Kg; SAD Cohort 4: ADEL Y-01 antibody at a dose of 50mg/Kg; SAD Cohort 5: ADEL Y-01 antibody at a dose of 100mg/Kg
Drug: Placebo - Healthy Participants — In Part 1 of our trial, we will enroll 2 placebo participants per cohort in up to 5 cohorts, undergoing the same protocol as those receiving ADEL-Y01 but with a placebo. They'll be part of the study from Day -1 to Day 4 for initial assessments and continue for 12 weeks for further safety and PK evaluations. This inclusion of placebo groups ensures a blinded study design for unbiased comparison of ADEL-Y01's safety and efficacy.
  Arms: SAD Cohort 1: Placebo at a dose of 2.5mg/Kg; SAD Cohort 2: Placebo at a dose of 7.5mg/Kg; SAD Cohort 3: Placebo at a dose of 20mg/Kg; SAD Cohort 4: Placebo at a dose of 50mg/Kg; SAD Cohort 5: Placebo at a dose of 100mg/Kg
Drug: ADEL-Y01 - MCI/AD — In Part 2 of our trial, we assess ADEL-Y01 in 33 participants aged 50 to 80 with MCI or mild AD, administering multiple IV doses every 2 weeks for 12 weeks. Each of the 3 cohorts will have 8 participants receiving ADEL-Y01, totaling 6 doses. After initial screening and consent, participants are randomized to start treatment on Day 1, with a follow-up in the clinical research unit for safety assessments. Additional safety and PK assessments occur bi-weekly up to 22 weeks, based on the start from the last dose on Day 71.
  Doses are set at 7.5, 20, and 50 mg/kg, adjusted based on Part 1 results and SRC safety reviews after at least 3 doses over 6 weeks. This phase focuses on understanding ADEL-Y01's safety and efficacy in AD patients through a cautious dosing strategy.
  Arms: MAD Cohort 1: ADEL Y-01 antibody at a dose of 7.5mg/Kg; MAD Cohort 2: ADEL Y-01 antibody at a dose of 20mg/Kg; MAD Cohort 3: ADEL Y-01 antibody at a dose of 50mg/Kg
Drug: Placebo - MCI/AD — In Part 2 of our clinical trial focusing on patients with MCI or mild AD, alongside the active treatment groups, we plan to include placebo groups within the 3 cohorts. Out of the 33 participants aged 50 to 80, 3 in each cohort, totaling 9 participants, will receive a placebo instead of the active drug, ADEL-Y01, administered every 2 weeks for 12 weeks. These placebo participants undergo the same screening, consent, and randomization procedures as those receiving the active drug. They are administered the placebo following the same schedule as the active groups, ensuring a controlled and blinded study environment to accurately assess ADEL-Y01's effects without bias.
  Placebo participants are crucial for comparing the active drug's impact on safety, tolerability, and effectiveness against a non-therapeutic intervention, maintaining the study's integrity and providing a benchmark for evaluating ADEL-Y01's true pharmacological effects on MCI or mild AD conditions.
  Arms: MAD Cohort 1: Placebo at a dose of 7.5mg/Kg; MAD Cohort 2: Placebo at a dose of 20mg/Kg; MAD Cohort 3: Placebo at a dose of 50mg/Kg

SUMMARY:
This is a Phase Ia/Ib, two-part, randomized, placebo-controlled, double-blinded, first in human(FIH) study to evaluate the safety, tolerability, PK, and PD of ADEL-Y01 in healthy participants in Part 1 and participants with MCI due to AD and mild AD in Part 2. The study includes 2 parts: Part 1 (single ascending dose [SAD] and Part 2 (multiple ascending dose [MAD]).

DETAILED DESCRIPTION:
The current standard of care (SoC) for Alzheimer's disease (AD) is aimed at improving memory and alertness only. There is an unmet medical need for an effective clinical treatment of neurodegeneration of AD and related dementia. Adel, Inc. and Oscotec Inc. are jointly developing a novel disease modifying immunotherapy agent (ADEL-Y01) targeting tubulin associated unit (tau) protein accumulation in the brain. ADEL-Y01 is a recombinant IgG1 class type monoclonal humanized antibody that recognizes and binds to tau protein acetylated at lysine-280 (K280) thus inhibiting aggregation and propagation of tau seeds and enhancing of microglial tau clearance. Administration of ADEL-Y01 has ameliorated memory impairment, behavioral deficits, and pathology in preclinical models. This first-in-human (FIH) study will assess the single and multiple dose safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD) of ADEL-Y01 in healthy adult participants and participants with mild cognitive impairment (MCI) due to AD and mild AD.

Part 1 (SAD): Part 1 will recruit up to 40 healthy participants, age 18 to 65 years inclusive. Up to 5 cohorts of 8 participants (6 active and 2 placebo participants per cohort) will be enrolled with each participant receiving ADEL-Y01 or placebo. Participants will be screened within 28 days of dose administration. The participants who will meet the inclusion/exclusion criteria for the study will be enrolled into the study after providing the informed consent form (ICF). The eligible participants will be randomized on Day -1 to receive either single dose of ADEL-Y01 or placebo on Day 1. Participants will be admitted on Day -1 and remain in the clinical research unit for at least 4 days (Day 4) following completion of all schedule procedures. Participants will return to the clinical research unit for additional safety and PK assessments on 7 occasions over a total of 12-weeks. Each dose level will include 2 sentinel participants (1 active and 1 placebo) who will be dosed first and monitored by the Investigator for at least 24 hours to check safety and tolerability. Once the safety of the study intervention is ensured, remaining participants will be dosed (5 active and 1 placebo). The starting dose for the Part 1 (SAD) will be 2.5 mg/kg. Subsequent dose levels are tentatively assigned to be 7.5, 20, 50 and 100 mg/kg. Dose escalation to the next dose level(s) will not proceed until the safety and tolerability of ADEL-Y01 results over an at least 14-day assessment period have been evaluated by the Safety Review Committee (SRC). A randomization list will be prepared for each cohort separately. No participant will be dosed more than once.

Part 2 (MAD): Part 2 will evaluate multiple IV doses of ADEL-Y01 administered every 2 weeks (Q2W) for 12 weeks in participants with MCI due to AD or mild AD. Thirty-three participants aged 50 to 80 years will be enrolled into 3 cohorts of 11 participants per cohort (8 active, 3 placebo) with each participant assigned to receive 6 doses of either ADEL-Y01 or placebo. Participants will be screened within 28 days of dose administration. The participants who will meet the inclusion/exclusion criteria for the study will be enrolled into the study after providing the ICF. The eligible participants will be randomized on Day -1 to receive either single dose of ADEL-Y01 or placebo on Day 1. Participants will be admitted on Day -1 and remain in the clinical research unit for at least 24 hours post infusion (Day 2) following completion of all schedule procedures. Participants will return to the clinical research unit for ADEL-Y01/placebo administration and/or additional safety and PK assessments on 12 occasions over a total of up to 22 weeks (ie, 12-weeks relative to the administration of the last dose of study intervention scheduled on Day 71). The provisional doses planned in Part 2 (MAD) are 7.5, 20, and 50 mg/kg administered every 2 weeks. The starting dose for the MAD part will be based on both safety and PK results from the Part 1 (SAD). The starting dose will be selected so that anticipated repeated-dose exposure to ADEL-Y01 (Cmax and AUC) does not exceed the exposure at the highest dose determined to be safe and well tolerated in the SAD. Depending on the Q2W ADEL-Y01 dose selected, the Part 2 (MAD) may commence prior to completion of the SAD study part. Dose escalation to the next dose level(s) will not proceed until the safety and tolerability of ADEL-Y01 over an at least 6-week assessment period (3 doses) have been evaluated by the SRC.

ELIGIBILITY:
Inclusion Criteria

Part 1: Participants are eligible to be included in the study only if all of the following criteria apply

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and/or female (of nonchildbearing potential) participants aged 18 to 65 years, inclusive.
3. A body mass index (BMI) between 18 to 30 kg/m2, inclusive.
4. Females must have a negative pregnancy test at the Screening Visit and on admission to the study center, must not be lactating and must be of nonchildbearing potential, confirmed at the Screening Visit by fulfilling 1 of the following criteria:

   * Postmenopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and with follicle stimulating hormone levels in the laboratory defined postmenopausal range.
   * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
5. Male participants should be willing to use double barrier contraception ie., condoms and spermicide, from the day of dosing until at least 3 months after dosing with the investigational product.
6. Male participant must not donate sperm from the day of dosing until at least 3 months after dosing with the investigational product.
7. Medically healthy with clinically insignificant screening results (eg, laboratory profiles, medical history, electrocardiograms [ECGs], and physical examination) as judged by the Principal Investigator.
8. Has to agree to abstain from alcohol intake 48 hours before administration of the study intervention and through the follow-up visit.
9. Able to be compliant with the protocol and attend all scheduled visits.

Part 2: Participants are eligible to be included in the study only if all of the following criteria apply

1. Age between 50 and 80 years.
2. Participants with MCI due to AD:

   i. Meet the National Institute on Aging - Alzheimer's Association (NIA-AA)6 core for MCI due to AD-intermediate likelihood.

   ii. Have a global clinical dementia rating (CDR) score of 0.5 and a CDR Memory Box score of 0.5 or greater at Screening and Baseline.

   iii. Report a history of subjective memory decline with gradual onset and slow progression over the last 1 year before Screening; must be corroborated by an informant.

   Participants with Mild AD dementia:

   iv. Meet the NIA-AA6 core for probable AD dementia. v. Have a global CDR score of 0.5 to 1.0 and a CDR Memory Box score of 0.5 or greater at Screening and Baseline.
3. Body weight of ≥50 kilograms and BMI between 18 and 35 kg/m2, inclusive.
4. Mini-Mental State Examination (MMSE) score of greater than or equal to 21 and less than or equal to 27 at screening.
5. Must have a positive amyloid positron emission tomography (within 12 months prior to screening) or CSF Abeta (42/40) ratio consistent with AD pathology.
6. Stable dose of AD treatment (Cholinesterase inhibitors [donepezil, rivastigmine, galantamine] and N-methyl-D-aspartate receptor antagonist [memantine]) 3 months before screening visit or being untreated.
7. Written informed consent must be obtained by participant or surrogate consenter (legally authorized representative).
8. Adequate visual and auditory abilities and language skills to allow neuropsychological testing.
9. Must be ambulatory.
10. Availability of partner/caregiver who spends at least 5 hours per week with the participant and is willing to act as a study partner and to consent for the study.
11. Participant on stable doses of all medications for concomitant illnesses according to medical history for at least 30 days prior to Visit 1 if considered relevant by the investigator.
12. Sexually active males and female must be using reliable contraception methods or be surgically sterile.

Exclusion Criteria

Part 1: Participants will be excluded from the study if any of the following criteria apply

1. History of any clinically important disease or disorder (major medical illnesses like cancer within 5 years, unstable angina or recent myocardial infarction, and renal failure) which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any current active infections, including localized infections, or any recent history (within 1 week prior to study intervention administration) of active infections (including severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2], cough or fever, or a history of recurrent or chronic infections).
4. Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational product or planned surgical procedure during the study period.
5. Any positive result at the Screening Visit for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus.
6. Blood donation within 1 month of screening or any blood donation/blood loss greater than 500 mL during the 3 months prior to screening.
7. Abnormal vital signs, after 10 minute supine rest at the Screening Visit and on Day -1, defined as any of the following:

   * Systolic blood pressure >140 mmHg.
   * Diastolic blood pressure >90 mmHg.
   * Heart rate <40 or >85 bpm.
8. Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG, and any clinically important abnormalities in the 12-lead ECG as considered by the Investigator that may interfere with the interpretation of QTc interval changes.
9. Prolonged Fridericia QT correction formula (QTcF) >450 msec at the Screening Visit and on Day -1.
10. Current smokers, or those who have smoked or used nicotine products within the previous 1 month.
11. History of alcohol abuse or excessive intake of alcohol defined as: an average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits.
12. Positive screen for alcohol, drugs of abuse or cotinine (≥400 ng/mL) at the Screening Visit or admission to the study center or positive screen for alcohol on admission to the study center prior to the first administration of investigational product.
13. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to any components in the investigational product.
14. Excessive intake of caffeine containing drinks or food eg, coffee, tea, chocolate, Red Bull, or cola (more than 6 cups of coffee or equivalent per day) within 7 days of investigational product administration. One caffeine unit is contained in the following items: 1 (6 oz) cup of coffee, 2 (12 oz) cans of cola, 1 (12 oz) cup of tea, ½ (4 oz) cup of energy drink (eg, Red Bull), or 3 (1 oz) chocolate bars.
15. Treatment with medications (including over-the-counter [OTC] medications, supplements, and herbal preparations such as St. John's Wort extract) within 14 days or 5 half-lives of the drug (whichever is longer) prior to investigational product administration, with the exception of a limited amount of acetaminophen (up to 2 g in 24 hours, but <1 g in 4 hours), which may be used throughout the study.
16. Has received another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment within at least minimum 3 months of the administration of investigational product in this study. The period of exclusion begins 3 months after the final dose (or greater than 5 times half-life) or 1 month after the last visit, whichever is the longest.

    Note: Participants consented and screened, but not dosed in this study or a previous Phase 1 study, are not excluded.
17. Ingestion of any poppy seeds within 24 hours. prior to each Drug Abuse Screening (Screening Visit and on Day -1 at check-in).
18. Previous randomization to treatment in the present study.
19. Involvement in the planning and/or conduct of the study (applies to the Sponsor, contract research organizations, and study center staff, etc.).
20. Participants who are unlikely to cooperate with the requirements of the study.
21. Judgment by the Investigator that the participant should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
22. Males with female partners of childbearing potential who are unwilling to use double barrier method of contraception for the duration of the study.

Part 2: Participants will be excluded from the study if any of the following criteria apply

1. History of any clinically important disease or disorder (major medical illnesses like cancer within 5 years, unstable angina or recent myocardial infarction, and renal failure) which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any positive result at the Screening Visit for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus.
4. Any current active infections, including localized infections, or any recent history (within 1 week prior to study intervention administration) of active infections (including SARS-CoV-2, cough or fever, or a history of recurrent or chronic infections).
5. Pregnant women.
6. Participation in another clinical study within 3 months before Visit 1.
7. Any medical or neurological condition other than AD that in the opinion of the investigator could be a contributing cause of the participant's dementia (eg, medication use, vitamin B12 deficiency, abnormal thyroid function, stroke or other cerebrovascular condition, diffuse Lewy body disease, head trauma).
8. History within the past 6 months or evidence of clinically significant psychiatric illness (eg, major depression, schizophrenia, or bipolar affective disorder).
9. Diagnosis of a dementia-related central nervous system disease other than AD (eg, Parkinson's Disease, Huntington's Disease, frontotemporal dementia, multi-infarct dementia, dementia with Lewy bodies, normal pressure hydrocephalus).
10. Identification of other known cause of dementia or any other clinically significant contributing co-morbid pathologies at screening magnetic resonance imaging (MRI), in the opinion of the investigator.
11. Participation in any other drug, biologic, device, or clinical study or treatment with any investigational drug or approved therapy for investigational use within 30 days (or 5 half-lives, whichever is longer) prior to screening, and/or participation in any other clinical study involving experimental medications for AD within 6 months (or 5 halflives, whichever is longer) prior to screening.
12. History and/or presence of autoimmune disease, if considered relevant by the investigator.
13. Contraindication for MRI such as MRI-incompatible metallic endoprosthesis or MRI incompatible stent implantation.
14. History of drug-induced cognitive impairment by benzodiazepines, strong sleeping aids, antipsychotics, narcotics, pain medicines like hydrocodone.
15. Participation in treatment with Lecanemab or any other disease modifying anti-amyloid drug.
16. History of alcohol abuse or excessive intake of alcohol defined as: an average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces(150 mL) of wine or 12 ounces(360 mL) of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits.
17. Positive screen for alcohol, drugs of abuse or cotinine (≥400 ng/mL) at the Screening Visit or admission to the study center or positive screen for alcohol on admission to the study center prior to the first administration of investigational product. A positive result for drugs of abuse is acceptable provided it can be linked a physician approved therapy.
18. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity to drugs likely to be used for this population, as judged by the Investigator or history of hypersensitivity to any components in the investigational product.
19. Ingestion of any poppy seeds within 24-hour prior to each drug abuse screening (Screening Visit and on Day -1 at check-in).
20. Previous randomization to treatment in the present study.
21. Involvement in the planning and/or conduct of the study (applies to the Sponsor, contract research organizations, and study center staff, etc.).
22. Participants who are unlikely to cooperate with the requirements of the study.
23. Judgment by the Investigator that the participant should not participate in the study if they have any ongoing or recent (ie, during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Evaluation of the safety and tolerability of ADEL-Y01 via single IV injection | D-28 ~ Week 12
  The standard safety and tolerability parameters to be assessed in the study include, but are not limited to, the following:
  Adverse Events (AEs) Vital signs, including blood pressure, pulse rate, pulse oximetry, respiratory rate, and body temperature Digital 12-lead ECGs Clinical laboratory assessments, encompassing hematology, biochemistry, coagulation, and urinalysis Physical examinations, which will include neurological assessments.
Part 2: Assessment of safety and tolerability with multiple IV Administrations of ADEL-Y01 in participants with MCI due to AD or Mild AD | D-28 ~ Week 22
  The study will assess standard safety and tolerability parameters, including but not limited to the following:
  Adverse Events (AEs) Vital signs such as blood pressure, pulse rate, pulse oximetry, respiratory rate, and body temperature Digital 12-lead ECGs Clinical laboratory assessments, including Hematology, Biochemistry, Coagulation, and Urinalysis Physical examinations, which will encompass neurological assessments C-SSRS (Columbia-Suicide Severity Rating Scale) assessments.

SECONDARY OUTCOMES:
Part 1: Characterization of the pharmacokinetics of ADEL-Y01 following a single IV injection | D-28 ~ Week 12
  The parameters and assessments in the study include serum Cmax, CEOI, tmax, AUC(0-last), AUC(0-inf), t1/2, λz, CL, Vss, Vz, as well as the incidence of anti-ADEL-Y01 antibodies in serum, ADEL-Y01 concentration at two specified time points (Day 2 and Day 15) in at least one cohort (20 mg/kg), and CSF to serum concentration ratios.
Part 1: Assessment of the immunogenicity of ADEL-Y01 following a single IV injection | D-28 ~ Week 12
  The parameters and assessments in the study include serum Cmax, CEOI, tmax, AUC(0-last), AUC(0-inf), t1/2, λz, CL, Vss, Vz, as well as the incidence of anti-ADEL-Y01 antibodies in serum, ADEL-Y01 concentration at two specified time points (Day 2 and Day 15) in at least one cohort (20 mg/kg), and CSF to serum concentration ratios.
Part 1: Assessment of the exposure to ADEL-Y01 in CSF following a single IV injection | D-28 ~ Week 12
  The parameters and assessments in the study include serum Cmax, CEOI, tmax, AUC(0-last), AUC(0-inf), t1/2, λz, CL, Vss, Vz, as well as the incidence of anti-ADEL-Y01 antibodies in serum, ADEL-Y01 concentration at two specified time points (Day 2 and Day 15) in at least one cohort (20 mg/kg), and CSF to serum concentration ratios.
Part 2: Characterization of the pharmacokinetics of ADEL-Y01 in participants with MCI due to AD and mild AD following multiple IV injections | D-28 ~ Week 22
  Assessing serum Cmax, tmax, AUC(0-last), AUC(0-tau), t1/2, CL, Vss, Vz, accumulation, and serum trough concentrations.
  Monitoring the incidence of anti-ADEL-Y01 antibodies in serum.
  Measuring CSF ADEL-Y01 concentration at two specified time points (1 day and 14 days after the final dose) from all cohorts, including CSF to serum concentration ratios.
  Evaluating changes in global function from baseline using the CDR-SB (Clinical Dementia Rating Scale Sum of Boxes) in participants with Alzheimer's disease.
  Assessing changes in cognitive function from baseline using the MMSE (Mini-Mental State Examination) in participants with Alzheimer's disease.
Part 2: Assessment of the immunogenicity of ADEL-Y01 in participants with MCI due to AD and mild AD following multiple IV injections | D-28 ~ Week 22
  Assessing serum Cmax, tmax, AUC(0-last), AUC(0-tau), t1/2, CL, Vss, Vz, accumulation, and serum trough concentrations.
  Monitoring the incidence of anti-ADEL-Y01 antibodies in serum.
  Measuring CSF ADEL-Y01 concentration at two specified time points (1 day and 14 days after the final dose) from all cohorts, including CSF to serum concentration ratios.
  Evaluating changes in global function from baseline using the CDR-SB (Clinical Dementia Rating Scale Sum of Boxes) in participants with Alzheimer's disease.
  Assessing changes in cognitive function from baseline using the MMSE (Mini-Mental State Examination) in participants with Alzheimer's disease.
Part 2: Assessment of the exposure to ADEL-Y01 in CSF in participants with MCI due to AD and mild AD following multiple IV injections. | D-28 ~ Week 22
  Assessing serum Cmax, tmax, AUC(0-last), AUC(0-tau), t1/2, CL, Vss, Vz, accumulation, and serum trough concentrations.
  Monitoring the incidence of anti-ADEL-Y01 antibodies in serum.
  Measuring CSF ADEL-Y01 concentration at two specified time points (1 day and 14 days after the final dose) from all cohorts, including CSF to serum concentration ratios.
  Evaluating changes in global function from baseline using the CDR-SB (Clinical Dementia Rating Scale Sum of Boxes) in participants with Alzheimer's disease.
  Assessing changes in cognitive function from baseline using the MMSE (Mini-Mental State Examination) in participants with Alzheimer's disease.
Part 2: Assessment of the preliminary clinical activity of ADEL-Y01 in participants with MCI due to AD and mild AD following multiple IV injections. | D-28 ~ Week 22
  Assessing serum Cmax, tmax, AUC(0-last), AUC(0-tau), t1/2, CL, Vss, Vz, accumulation, and serum trough concentrations.
  Monitoring the incidence of anti-ADEL-Y01 antibodies in serum.
  Measuring CSF ADEL-Y01 concentration at two specified time points (1 day and 14 days after the final dose) from all cohorts, including CSF to serum concentration ratios.
  Evaluating changes in global function from baseline using the CDR-SB (Clinical Dementia Rating Scale Sum of Boxes) in participants with Alzheimer's disease.
  Assessing changes in cognitive function from baseline using the MMSE (Mini-Mental State Examination) in participants with Alzheimer's disease.

OTHER OUTCOMES:
Assessment of ADEL-Y01 Effects on Biomarkers in CSF and Plasma in Participants with MCI due to AD and Mild AD for Exploratory Objective | D-28 ~ Week 22
  Collection of blood and CSF samples for biomarker research will be performed in Part 2 of the study. Samples will be tested for potential biomarkers in CSF, plasma and/or serum to evaluate PD changes with exposure to ADEL-Y01 and their association with the observed clinical responses to ADEL-Y01. The following samples (CSF and/or blood) for biomarker research will be collected from all participants in this study. Analysis may be performed on biomarker variants thought to play a role in tauopathy in AD to evaluate their association with observed clinical responses to ADEL-Y01 administration. Biomarkers to be tested include, but are not limited to, the following: Aβ1-40, Aβ1-42, p-tau217, t-tau, acK280Tau, MTBR243, and others (for example, neurodegeneration/inflammation multiplex assay including NfL, GFAP, YKL-40, and biomarkers determined by proteomic analysis such as OLINK Proteomic Microassay).

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Yong Yoon, Study Chair — Alzheimer's Disease Expert Lab (ADEL), Inc.
Locations (6):
- United States (6):
  - CenExel ACT, Anaheim, California
  - K2 Medical Research - The Villages, Lady Lake, Florida
  - K2 Medical Research - Orlando, Maitland, Florida
  - Innovation Medical Research, Palmetto Bay, Florida
  - Accel Research - Neurostudies, Decatur, Georgia
  - Quest Research Institute, Farmington Hills, Michigan

IPD SHARING:
Plan to Share IPD: Undecided
We intend to provide future updates that prioritize transparency in sharing results.